CLINICAL TRIAL: NCT00002337
Title: A Phase I Safety and Tolerability Study of Four Doses of OPC-8212 (Vesnarinone) in Advanced HIV Disease
Brief Title: A Study of Multiple Doses of Vesnarinone in Advanced HIV Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 234B; 22-93-252
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antiviral Agents; vesnarinone
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vesnarinone

INTERVENTIONS:
Drug: Vesnarinone

SUMMARY:
To evaluate the safety and tolerability of four doses of oral vesnarinone in patients with advanced HIV disease.

DETAILED DESCRIPTION:
Fourteen patients per dose level receive vesnarinone at 1 of 4 doses for 12 weeks. At least seven patients at a given dose level must have completed 4 weeks of treatment before dose is escalated in subsequent patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii, candida, mycobacteria, and other opportunistic infections.
* Acyclovir for up to 14 days for acute herpes outbreaks.

Patients must have:

* Documented HIV infection.
* CD4 count 50 - 300 cells/mm3.
* No active opportunistic infections.
* No fever, diarrhea, or Herpes zoster.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant current cardiac disease, including patients who exhibit long QTC syndrome on EKG screening and who have an abnormal cardiothoracic ratio on chest x-ray at baseline.
* Active malignancy (other than cutaneous Kaposi's sarcoma or cutaneous basal cell carcinoma or in situ carcinoma of the cervix).

Concurrent Medication:

Excluded:

* Antiretroviral agents, including ddI, ddC, AZT, and d4T.
* Immunosuppressive agents.
* Investigational HIV drugs/therapies including vaccines.
* Interferon or other immunomodulating agents.
* Corticosteroids (other than topical).
* Hematopoietins.
* Megestrol acetate.
* Agents known to cause neutropenia.
* Trimethoprim/sulfamethoxazole in excess of 160 mg trimethoprim and 800 mg sulfamethoxazole thrice weekly.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* Prior history of cardiac disease.
* History of agranulocytosis or severe (grade 3 or worse) drug-induced neutropenia or documented abnormalities in granulocyte function.

Prior Medication:

Excluded:

* AZT, ddI, ddC, d4T, or other nucleoside analog antiretroviral therapy within 14 days prior to study entry.
* Prior cytotoxic chemotherapy.
* Acyclovir for herpes prophylaxis within 48 hours prior to study entry.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Erythropoietin, transfusion, or blood product use.
* Radiation therapy (including electron beam irradiation). Active use of illicit drugs (specifically cocaine, amyl nitrate, heroin, and other cardioactive agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56

CONTACTS AND LOCATIONS:
Locations (1):
- AIDS Research Consortium of Atlanta, Atlanta, Georgia, United States